CLINICAL TRIAL: NCT04791917
Title: Marijuana Use, Strength Training, and Alcohol Consumption (MUSTAC) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Research Society on Alcohol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202000058-N; 1F31AA028696-01A1 (NIH); AGR DTD 02-17-2020 (Other Grant/Funding Number: Research Society on Alcoholism); UFCAREDAG002 (Other Grant/Funding Number: UF Center for Addiction Research and Education); 00045887 (Other Grant/Funding Number: UF Dept of Clinical and Health Psychology)
Record Dates: First submitted 2021-03-09; First posted 2021-03-10 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Onset Muscle Soreness Induction (Experimental): Participants will complete an exercise session designed to induce delayed onset muscle soreness in the biceps
  Interventions: Behavioral: Eccentric Biceps Flexion
- Sham Delayed Onset Muscle Soreness Induction (Sham Comparator): Participants will complete an exercise session that is unlikely to induce delayed onset muscle soreness in the biceps
  Interventions: Behavioral: Concentric Biceps Flexion

INTERVENTIONS:
Behavioral: Eccentric Biceps Flexion — Muscle lengthening biceps exercise
  Arms: Delayed Onset Muscle Soreness Induction
Behavioral: Concentric Biceps Flexion — Muscle shortening biceps exercise
  Arms: Sham Delayed Onset Muscle Soreness Induction

SUMMARY:
Self-medication of pain by consuming alcohol and marijuana is common. However, the research regarding pain as a determinant for alcohol and marijuana use has relied on laboratory pain induction paradigms with limited clinical relevance. The study will assess demand for alcohol and marijuana before and after delayed onset muscle soreness (DOMS) induction in co-users. This will provide a clinically relevant, but time-limited, model for the effects of musculoskeletal pain on demand.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years;
* English-speaking
* Self-identify as White/Caucasian or Black/African American
* Own a smartphone with cellular/data plan
* Regularly co-use alcohol and smoked marijuana as indicated by scores of ≥3 on item 1 of the CUDIT-R and AUDIT.
* Willing and able to give informed consent

Exclusion Criteria:

* Participation in biceps-specific conditioning program in the past 6 months*
* Self-reported wrist/hand, elbow, or shoulder pain the past 3 months
* Chronic medical condition that may affect pain perception (e.g. diabetes, fibromyalgia, headaches)
* Self-reported kidney dysfunction, muscle damage, or major psychiatric disorder
* Medical marijuana prescription
* Consumption of marijuana using only non-inhalational methods (e.g. edibles, tinctures, or cannabidiol oil)
* Score of ≥ 10 on Patient Health Questionnaire-9 (moderate depression)
* Women who are pregnant, trying to become pregnant, or breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Boissoneault, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Center for Pain Research and Behavioral Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delayed Onset Muscle Soreness Induction | Sham Delayed Onset Muscle Soreness Induction
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Onset Muscle Soreness Induction | Sham Delayed Onset Muscle Soreness Induction | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.77 (7.46) | 29.48 (11.81) | 27.08 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 51
Employment [Count of Participants; unit: Participants]
  Employed | 14 | 10 | 24
  Unemployed | 12 | 15 | 27
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-9 (PHQ-9). Measure of depressive symptomatology over the past 2 weeks. Scores range from 0-27, with higher scores reflecting more severe depression.
  units on a scale | 4.35 (3.17) | 4.92 (4.34) | 4.63 (3.76)
GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder-7 (GAD-7) questionnaire. Measures anxiety over the last 2 weeks. Scores range from 0-21, with higher scores reflecting more severe anxiety.
  units on a scale | 5.00 (4.52) | 4.12 (3.43) | 4.57 (4.01)
Alcohol Use Urge [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing current urge to consume alcohol, anchored from 'no urge' to 'very strong urge'. Scores range from 0-100, with higher scores reflecting stronger urge.
  visual analog scale units | 19.96 (24.51) | 40.64 (28.05) | 29.44 (27.92)
Cannabis Use Urge [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing current urge to consume cannabis, anchored from 'no urge' to 'very strong urge'. Scores range from 0-100, with higher scores reflecting stronger urge.
  visual analog scale units | 44.81 (34.02) | 67.58 (23.99) | 55.74 (31.51)
Pain-related Negative Affect [Mean (Standard Deviation); unit: total score] — Sum of responses to 0-100 visual analog scales (VASs) assessing current depression, anxiety, frustration, fear, and anger anchored from 'none' to 'worst imaginable'. Total scores range from 0-500, with higher scores reflecting greater pain-related negative affect.
  total score | 139.46 (90.40) | 140.36 (103.37) | 139.90 (96.00)
Negative Urgency [Mean (Standard Deviation); unit: units on UPPS-P subscale] — Negative Urgency subscale of the short form of the Urgency, Premeditation, Perseverance, Sensation Seeking, Positive Urgency, Impulsive Behavior Scale (UPPS-P). Scores are sums of reverse coded responses to items 6, 8, 13, and 15 and range from 0-12, with higher scores reflecting greater negative urgency.
  units on UPPS-P subscale | 8.35 (2.95) | 8.67 (2.82) | 8.50 (2.87)
History of Alcohol Self-Medication [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing frequency of alcohol use in the past to cope with pain, anchored from 'none of the time' to 'all of the time'. Scores range from 0-100, with higher scores reflecting more frequent self-medication.
  visual analog scale units | 57.28 (54.59) | 73.96 (45.19) | 65.62 (50.31)
History of Cannabis Self-Medication [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing frequency of cannabis use in the past to cope with pain, anchored from 'none of the time' to 'all of the time'. Scores range from 0-100, with higher scores reflecting more frequent self-medication.
  visual analog scale units | 107.31 (60.77) | 114.08 (58.64) | 110.63 (59.24)
Alcohol Expectancy VAS 1 [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing belief that using alcohol would provide relief from pain, anchored from 'no pain relief at all' to 'complete pain relief'. Scores range from 0-100, with higher scores reflecting stronger belief that alcohol use will relieve pain.
  visual analog scale units | 37.08 (29.29) | 44.72 (26.33) | 40.90 (27.83)
Alcohol Expectancy VAS 2 [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing belief that using alcohol would affect pain sensitivity, anchored from 'strongly decreased' to 'strongly increased'. Scores range from 0-100, with higher scores reflecting stronger belief that alcohol use will increase pain sensitivity.
  visual analog scale units | 25.81 (18.31) | 28.20 (16.89) | 26.98 (17.53)
Cannabis Expectancy VAS 1 [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing belief that using cannabis would provide relief from pain, anchored from 'no pain relief at all' to 'complete pain relief'. Scores range from 0-100, with higher scores reflecting stronger belief that cannabis use will relieve pain.
  visual analog scale units | 62.35 (28.27) | 71.76 (18.82) | 66.96 (24.34)
Cannabis Expectancy VAS 2 [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing belief that using cannabis would affect pain sensitivity, anchored from 'strongly decreased' to 'strongly increased'. Scores range from 0-100, with higher scores reflecting stronger belief that cannabis use will increase pain sensitivity.
  visual analog scale units | 38.32 (26.93) | 38.08 (26.71) | 38.20 (26.54)
AUDIT Total Score [Mean (Standard Deviation); unit: units on a scale] — Total score on the Alcohol Use Disorders Identification Test (AUDIT), which assesses alcohol use disorder symptomatology. Scores range from 0-40, with higher scores indicating more severe symptomatology.
  units on a scale | 10.54 (4.52) | 11.36 (5.99) | 10.94 (5.26)
CUDIT Total Score [Mean (Standard Deviation); unit: units on a scale] — Total score on the Cannabis Use Disorders Identification Test (CUDIT), which assesses cannabis use disorder symptomatology. Scores range from 0-40, with higher scores indicating more severe symptomatology.
  units on a scale | 11.77 (4.92) | 14.57 (7.12) | 13.14 (6.20)
ASSIST Cannabis Risk Score [Mean (Standard Deviation); unit: units on a scale] — Cannabis risk score derived from the World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), which assesses substance use-related health risks. Scores range from 0-42, with higher scores indicating higher risk.
  units on a scale | 13.62 (7.23) | 15.28 (6.57) | 14.43 (6.90)
Alcohol Use Frequency [Count of Participants; unit: Participants]
  2 to 3 times a week | 21 | 18 | 39
  4 or more times a week | 5 | 7 | 12
Drinks Per Drinking Day [Count of Participants; unit: Participants]
  1 or 2 | 7 | 11 | 18
  3 or 4 | 9 | 8 | 17
  5 or 6 | 8 | 4 | 12
  7 to 9 | 2 | 2 | 4
Cannabis Use Frequency [Count of Participants; unit: Participants]
  Once a week | 1 | 1 | 2
  Twice a week | 9 | 3 | 12
  3-4 times a week | 7 | 9 | 16
  5-6 times a week | 1 | 5 | 6
  Once a day | 4 | 2 | 6
  More than once a day | 4 | 5 | 9
Duration of Cannabis Use at Current Frequency [Count of Participants; unit: Participants]
  1-3 months | 3 | 2 | 5
  3-6 months | 2 | 2 | 4
  6-9 months | 1 | 2 | 3
  9-12 months | 3 | 0 | 3
  1-2 years | 7 | 6 | 13
  2-3 years | 5 | 2 | 7
  3-5 years | 1 | 5 | 6
  5-10 years | 3 | 2 | 5
  10-15 years | 1 | 1 | 2
  More than 20 years | 0 | 3 | 3
Primary Method Used to Ingest Cannabis [Count of Participants; unit: Participants]
  Joints | 6 | 10 | 16
  Blunts | 5 | 3 | 8
  Hand pipe | 6 | 4 | 10
  Bong/Water Pipe | 6 | 5 | 11
  Vaporizer | 3 | 1 | 4
  Edibles | 0 | 1 | 1
  Other | 0 | 1 | 1
Primary Form of Cannabis Used [Count of Participants; unit: Participants]
  Flower/Herbal Cannabis | 24 | 23 | 47
  Concentrates (e.g., oil, wax, shatter, hash, dabs) | 2 | 1 | 3
  Edibles | 0 | 1 | 1
Frequency of Simultaneous Alcohol and Cannabis Use [Mean (Standard Deviation); unit: visual analog scale units] — Visual analog scale (VAS) assessing frequency of simultaneous use of alcohol and cannabis over the past 12 months (such that effects overlapped), anchored from 'not at all' to 'every time'. Scores range from 0-100, with higher scores reflecting more frequent simultaneous use.
  visual analog scale units | 53 (19.17) | 62.32 (21.26) | 57.76 (20.60)
Amount Spent on Alcohol in Past Month [Mean (Standard Deviation); unit: dollars] | 84.77 (79.49) | 110.48 (84.08) | 97.33 (81.82)
Amount Spent on Cannabis in Past Month [Mean (Standard Deviation); unit: dollars] | 88.86 (90.10) | 102.62 (113.91) | 95.58 (101.43)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Demand: Breakpoint
Description: Changes in breakpoint of alcohol demand, assessed using the Alcohol Purchase Task. Breakpoint indicates the drink price at which participants report no alcohol consumption. Values represent difference scores derived from breakpoint values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: dollars/drink
Groups:
- Delayed Onset Muscle Soreness Induction (Women); Delayed Onset Muscle Soreness Induction (Men): Participants will complete an exercise session designed to induce delayed onset muscle soreness in the biceps
  Eccentric Biceps Flexion: Muscle lengthening biceps exercise
- Sham Delayed Onset Muscle Soreness Induction (Women); Sham Delayed Onset Muscle Soreness Induction (Men): Participants will complete an exercise session that is unlikely to induce delayed onset muscle soreness in the biceps
  Concentric Biceps Flexion: Muscle shortening biceps exercise
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
dollars/drink | -6.00 (7.62) | -2.07 (5.61) | -1.81 (4.45) | -1.09 (8.51)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on breakpoint for alcohol including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .26, ANCOVA; F(1,41) = 1.32, partial eta squared = .03

2. Primary Outcome: Alcohol Demand: Omax
Description: Changes in Omax, assessed using the Alcohol Purchase Task. Omax reflects the highest total amount in dollars that a participant would spend on alcohol-containing beverages. Values represent difference scores derived from log-transformed Omax values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: (log)dollars
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
(log)dollars | -.255 (.497) | -.089 (.20) | -.03 (.40) | -.168 (.36)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Omax for alcohol including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .11, ANCOVA; F(1,43) = 2.60, partial eta squared = .06

3. Primary Outcome: Alcohol Demand: Pmax
Description: Changes in Pmax, assessed using the Alcohol Purchase Task. Pmax reflects the price point at which demand for alcohol becomes elastic (i.e., declines in response to increasing price). Values represent difference scores derived from log-transformed Pmax values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: log(dollars/drink)
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
log(dollars/drink) | -.19 (.36) | -.080 (.24) | .0054 (.24) | -.11 (.299)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on alcohol Pmax including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .17, ANCOVA; F(1,42) = 1.95, partial eta squared = .04

4. Primary Outcome: Alcohol Demand: Essential Value
Description: Changes in Essential Value, assessed using the Alcohol Purchase Task. Essential Value represents the reinforcing efficacy of alcohol, such that higher Essential Value indicates greater reinforcing efficacy. Values represent difference scores derived from Essential Values coded so that positive numbers indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
index | -.18 (.25) | -.072 (.18) | -.24 (.22) | -.073 (.28)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on alcohol essential value including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .91, ANCOVA; F(1,43)=.01, partial eta squared = .00

5. Primary Outcome: Cannabis Demand: Intensity
Description: Changes in intensity of cannabis demand, assessed using the Marijuana Purchase Task. Intensity reflects the number of joints that would hypothetically be consumed if they were free. Values represent difference scores derived from log-transformed intensity values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: (log)joints
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
(log)joints | -.019 (.28) | .12 (.39) | -.070 (.31) | -.10 (.54)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on intensity of cannabis demand including baseline urge to consume cannabis and CUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .14, ANCOVA; F(1,41) = 2.24, partial eta squared = .05

6. Primary Outcome: Cannabis Demand: Breakpoint
Description: Changes in breakpoint of cannabis demand, assessed using the Marijuana Purchase Task. Breakpoint indicates the joint price at which participants report no cannabis consumption. Values represent difference scores derived from breakpoint values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: dollars/joint
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
dollars/joint | .40 (1.78) | -.14 (1.97) | -.36 (1.88) | -.80 (1.59)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on breakpoint of cannabis demand including baseline urge to consume cannabis and CUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .83, ANCOVA; F(1,41) = .04, partial eta squared = .001

7. Primary Outcome: Cannabis Demand: Omax
Description: Changes in Omax, assessed using the Marijuana Purchase Task. Omax reflects the highest total amount that a participant would spend on cannabis. Values represent difference scores derived from log-transformed Omax values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: (log)dollars
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
(log)dollars | .019 (.45) | -.010 (.20) | -.001 (.26) | -.10 (.40)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Omax for cannabis including baseline urge to consume cannabis and CUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .15, ANCOVA; F(1,41) = 2.20, partial eta squared = .05

8. Primary Outcome: Cannabis Demand: Pmax
Description: Changes in Pmax, assessed using the Marijuana Purchase Task. Pmax reflects the price point at which demand for cannabis becomes elastic (i.e., declines in response to increasing price). Values represent difference scores derived from log-transformed Pmax values coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: log(dollars/joint)
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
log(dollars/joint) | .0005 (.22) | -.043 (.21) | .014 (.24) | -.10 (.31)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .24, ANCOVA; F(1,41) = 1.41, partial eta squared = .03

9. Primary Outcome: Cannabis Demand: Essential Value
Description: Changes in Essential Value, assessed using the Marijuana Purchase Task. Essential Value represents the reinforcing efficacy of cannabis, such that higher Essential Value indicates greater reinforcing efficacy. Values represent difference scores derived from Essential Values coded so that positive numbers indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
index | -.061 (.23) | .059 (.23) | -.032 (.162) | .15 (.27)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Essential Value for cannabis including baseline urge to consume cannabis and CUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .97, ANCOVA; F(1,41) = .001, partial eta squared = .00
Statistical Analysis 2: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Essential Value for cannabis including baseline urge to consume cannabis and CUDIT score as covariates. Here we report the results of the analysis of the Time X Group interaction; Test type: Superiority; p = .03, ANCOVA; F(1,41) = 4.86, partial eta squared = .11

10. Primary Outcome: Alcohol Demand: Intensity
Description: Changes in intensity of alcohol demand, assessed using the Alcohol Purchase Task. Intensity reflects the number of drinks that would hypothetically be consumed if they were free. Values represent difference scores derived from log-transformed number of drinks coded so that positive values indicate an increase in the demand index from baseline to follow-up.
Time Frame: 48 hours after exercise
Measure: Mean (Standard Deviation); unit: log(drinks)
Arm/Group | Delayed Onset Muscle Soreness Induction (Women) | Sham Delayed Onset Muscle Soreness Induction (Women) | Delayed Onset Muscle Soreness Induction (Men) | Sham Delayed Onset Muscle Soreness Induction (Men)
Number analyzed (Participants) | 15 | 14 | 11 | 11
log(drinks) | -.094 (.295) | .047 (.15) | .0958 (.285) | -.07 (.33)
Statistical Analysis 1: Comparison: Delayed Onset Muscle Soreness Induction (Women) vs Sham Delayed Onset Muscle Soreness Induction (Women) vs Delayed Onset Muscle Soreness Induction (Men) vs Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on intensity of alcohol demand including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the Sex X Time X Group interaction; Test type: Superiority; p = .04, ANCOVA; F(1,42) = 4.66, partial eta squared = .10
Statistical Analysis 2: Comparison: Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Intensity of alcohol demand including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the effect of Time on Intensity for men in the DOMS group; Test type: Superiority; p = .26, ANCOVA; Slope = .10
Statistical Analysis 3: Comparison: Delayed Onset Muscle Soreness Induction (Women); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Intensity of alcohol demand including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the effect of Time on Intensity for women in the DOMS group; Test type: Superiority; p = .22, ANCOVA; Slope = -.09
Statistical Analysis 4: Comparison: Sham Delayed Onset Muscle Soreness Induction (Men); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Intensity of alcohol demand including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the effect of Time on Intensity for men in the sham DOMS group; Test type: Superiority; p = .27, ANCOVA; Slope = -.10
Statistical Analysis 5: Comparison: Sham Delayed Onset Muscle Soreness Induction (Women); 2 (Sex: men vs. women) X 2 (Time: Pre- vs. post-exercise) x 2 (Group: DOMS vs. sham DOMS) mixed general linear model on Intensity of alcohol demand including baseline urge to consume alcohol and AUDIT score as covariates. Here we report the results of the analysis of the effect of Time on Intensity for women in the sham DOMS group; Test type: Superiority; p = .49, ANCOVA; Slope = .06

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Delayed Onset Muscle Soreness Induction | Sham Delayed Onset Muscle Soreness Induction
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT04791917/Prot_SAP_ICF_000.pdf